CLINICAL TRIAL: NCT05875675
Title: Effect of Pioglitazone Treatment in Patient's Calcific Aortic Valve Disease With Mild Aortic Valve Stenosis
Brief Title: Effects of Pioglitazone in Calcific Aortic Valve Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WUHFACAVD02
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Calcification of Aortic Valve; Aortic Valve Stenosis
Keywords: Calcification of Aortic Valve; Aortic Valve Stenosis; Pioglitazone
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug group (Experimental): Dietary Supplement: Pioglitazone 30 mg by mouth daily
  Interventions: Drug: Drug: Pioglitazone Oral Tablet
- Control group (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Drug: Pioglitazone Oral Tablet — Dietary Supplement: Pioglitazone 30 mg by mouth daily
  Arms: Drug group
Dietary Supplement: Placebo — Dietary: Supplement: Placebo
  Arms: Control group

SUMMARY:
This is a prospective, randomized, comparative, clinical trial conducted by Wuhan Union Hospital that aims to evaluate the efficacy and safety of pioglitazone compared to placebo in patients with calcific aortic valve disease with mild aortic valve stenosis.

DETAILED DESCRIPTION:
Pioglitazone is an oral drug for the treatment of type 2 diabetes that improves the utilization of glucose by the body by inhibiting hepatic gluconeogenesis, and has anti-inflammatory and antioxidant effects that may improve vascular endothelial cell injury and prevent cardiovascular disease. This study is to slow the process of aortic valve calcification by pioglitazone intervention with the aim of reducing the risk of aortic valve stenosis. Participants were randomized into two groups: one group was given oral pioglitazone treatment and the other group was given placebo control. Patients in both groups were observed for aortic valve calcification during the follow-up period, and changes in aortic valve thickness, degree of calcification, and flow were recorded by cardiac ultrasonography, while the incidence of cardiovascular events and adverse effects were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 35 years of age at the time of rescruiting.
* Subject has calcific aortic valve disease with mild to moderate aortic valve stenosis as defined by Doppler echocardiography results: Aortic Valve mean pressure gradient between 10-30 mmHg and Aortic Valve Area ≥ 1.2 and ≤ 2.0 cm2 on TTE within 2 weeks prior to randomization and Cardiac Compute Tomography (CT) test results: aortic valve calcium score (Agatston score) ≥ 200 AU at baseline cardiac CT within 1 month prior to randomization
* Subject provides written informed consent prior to initiation of any study procedures.
* Subject understands and agrees to comply with planned study procedures.

Exclusion Criteria:

* Subject has concomitant moderate or severe mitral or tricuspid valve disease.
* Subject has left ventricular ejection fraction < 50%.
* Subject previous history of aortic valve surgery, pancreatitis, malignant tumor, drug or alcohol abuse.
* Subjects whose alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal range.
* Subjects who cannot undergo Cardiac CT.
* Pregnant or lactating women.
* Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  overall survival (OS)

SECONDARY OUTCOMES:
Time-to-major adverse cardiovascular events | 104 weeks
  Time-to-major adverse cardiovascular events of cardiac death, non- fatal myocardial infarction, heart failure hospitalization and stroke
Change in aortic valve stenosis severity | at week 104
  Change in aortic valve stenosis severity as measured by peak transaortic velocity using echocardiography at week 104 as compared to baseline
HbA1c | 104 weeks
  Metabolic control
Glucose level | 104 weeks
  Metabolic control

IPD SHARING:
Plan to Share IPD: Yes
we would like to share IPD with other researchers 1 years after the trial completely finished
Supporting Information: Study Protocol, ICF, CSR
Time Frame: All data should only be used for academic research.

REFERENCES:
- [Background] Chu Y, Lund DD, Weiss RM, Brooks RM, Doshi H, Hajj GP, Sigmund CD, Heistad DD. Pioglitazone attenuates valvular calcification induced by hypercholesterolemia. Arterioscler Thromb Vasc Biol. 2013 Mar;33(3):523-32. doi: 10.1161/ATVBAHA.112.300794. Epub 2013 Jan 3. PMID 23288158
- [Background] Greenberg HZE, Zhao G, Shah AM, Zhang M. Role of oxidative stress in calcific aortic valve disease and its therapeutic implications. Cardiovasc Res. 2022 May 6;118(6):1433-1451. doi: 10.1093/cvr/cvab142. PMID 33881501
- [Background] Hajj GP, Chu Y, Lund DD, Magida JA, Funk ND, Brooks RM, Baumbach GL, Zimmerman KA, Davis MK, El Accaoui RN, Hameed T, Doshi H, Chen B, Leinwand LA, Song LS, Heistad DD, Weiss RM. Spontaneous Aortic Regurgitation and Valvular Cardiomyopathy in Mice. Arterioscler Thromb Vasc Biol. 2015 Jul;35(7):1653-62. doi: 10.1161/ATVBAHA.115.305729. Epub 2015 May 21. PMID 25997932
- [Background] Weiss RM, Miller JD, Heistad DD. Fibrocalcific aortic valve disease: opportunity to understand disease mechanisms using mouse models. Circ Res. 2013 Jul 5;113(2):209-22. doi: 10.1161/CIRCRESAHA.113.300153. PMID 23833295